CLINICAL TRIAL: NCT01699737
Title: A Phase 2, Randomized, Double-blind, Double-dummy, Placebo and Active-controlled, Multicenter, Parallel Group Study to Evaluate the Efficacy and Safety of JTT-851 in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy Study of JTT-851 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT851-U-12-002
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — glimepiride; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- JTT-851 Dose 1 (Experimental): JTT-851 Tablets and Placebo comparator capsule, administered once daily for 12 weeks
  Interventions: Drug: JTT-851; Drug: Placebo for comparator
- JTT-851 Dose 2 (Experimental): JTT-851 Tablets and Placebo comparator capsule, administered once daily for 12 weeks
  Interventions: Drug: JTT-851; Drug: Placebo for comparator
- JTT-851 Dose 3 (Experimental): JTT-851 Tablets and Placebo comparator capsule, administered once daily for 12 weeks
  Interventions: Drug: JTT-851; Drug: Placebo for comparator
- Glimepiride Dose 1 (Active Comparator): Active Comparator Capsule and Placebo Tablets, administered once daily for 12 weeks
  Interventions: Drug: Glimepiride; Drug: Placebo for Active
- Placebo active & Placebo comparator (Placebo Comparator): Placebo Tablets for study drug and Placebo Capsule for active comparator, administered once daily for 12 weeks
  Interventions: Drug: Placebo for Active; Drug: Placebo for comparator

INTERVENTIONS:
Drug: JTT-851
  Arms: JTT-851 Dose 1; JTT-851 Dose 2; JTT-851 Dose 3
Drug: Glimepiride — Encapsulated Glimepiride tablets
  Arms: Glimepiride Dose 1
Drug: Placebo for Active
  Arms: Glimepiride Dose 1; Placebo active & Placebo comparator
Drug: Placebo for comparator
  Arms: JTT-851 Dose 1; JTT-851 Dose 2; JTT-851 Dose 3; Placebo active & Placebo comparator

SUMMARY:
The purpose of this study is to evaluate the effect of JTT-851 on diabetes as well as to assess the safety, tolerability, and pharmacokinetics of JTT-851 in type 2 diabetic patients either treated with metformin or treatment-naïve.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, placebo and active-controlled (glimepiride), multi-center, parallel-group study to investigate the effect of JTT-851 on HbA1c and other ancillary efficacy parameters and to assess the safety, tolerability, and pharmacokinetics of JTT-851 in inadequately-controlled treatment-naïve or metformin-treated type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with type 2 diabetes, 18-70 years of age at Visit 1
* Managing diabetes with diet and exercise only or currently being treated with a stable dose of metformin (at least 1500 mg/day)
* Glycosylated hemoglobin at Visit 1 between 7.5% and 10.0%, if on metformin and between 7.5% and 10.9%, if without treatment
* Body mass index (BMI) ≥ 23.0 kg/m^2 and ≤ 45.0 kg/m^2 at Visit 1

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* Known medical history or presence of type 1 diabetes or acute metabolic diabetic complications, unstable or rapidly progressing retinopathy, nephropathy or neuropathy
* Acute coronary syndrome or uncontrolled hypertension
* Does not meet all diet or previous/concomitant medication restriction criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c) after administration of JTT-851 | 12 weeks
  To investigate the change in glycosylated hemoglobin (HbA1c) after JTT-851 administration, once daily for 12 weeks

SECONDARY OUTCOMES:
Safety and tolerability of JTT-851 in patients with type 2 diabetes compared to glimepiride and placebo | 12 weeks
  To evaluate the safety and tolerability of JTT-851 when administered for 12 weeks in patients with type 2 diabetes compared to glimepiride and placebo.
Effect on ancillary efficacy measures | 12 weeks
  To investigate the effect of JTT-851 administration on ancillary efficacy measures in patients with type 2 diabetes compared to glimepiride and placebo.
Pharmacokinetics of JTT-851 and its metabolites | 12 weeks
  To evaluate the pharmacokinetics of JTT-851 and its metabolites in patients with type 2 diabetes

OTHER OUTCOMES:
Relationship between dose and response of JTT-851 | 12 weeks
  To explore the relationship between the JTT-851 dose (exposure) and response

CONTACTS AND LOCATIONS:
Overall Officials: Hisashi Kodama, Ph.D., Study Chair — Akros Pharma Inc.
Locations (79):
- United States (79):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Muscle Shoals, Alabama
  - Glendale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Artesia, California
  - Beverly Hills, California
  - Buena Park, California
  - Chino, California
  - Garden Grove, California
  - Lincoln, California
  - Lomita, California
  - Los Angeles, California
  - Newport Beach, California
  - North Hollywood, California
  - Paramount, California
  - Sacramento, California
  - Spring Valley, California
  - Walnut Creek, California
  - Denver, Colorado
  - Cooper City, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Kissimee, Florida
  - Miami, Florida
  - Miramar, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Columbus, Georgia
  - Marietta, Georgia
  - Nampa, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - New Orleans, Louisiana
  - Oxon Hill, Maryland
  - Olive Branch, Mississippi
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Mine Hill, New Jersey
  - Glen Falls, New York
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Marion, Ohio
  - Munroe Falls, Ohio
  - Wadsworth, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Lansdale, Pennsylvania
  - Columbia, South Carolina
  - Greer, South Carolina
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Sugarland, Texas
  - Tomball, Texas
  - Murray, Utah
  - Orem, Utah
  - Salt Lake City, Utah
  - Burke, Virginia
  - Manassas, Virginia
  - Norfolk, Virginia
  - Suffolk, Virginia
  - Madison, Wisconsin